CLINICAL TRIAL: NCT00249704
Title: Evaluation of the Effect of a 4-Month Intervention of Exercise and/or Vitamin D on Mobility Function and Strength in Frail Elderly Subjects
Brief Title: Randomized Study Of Exercise And Vitamin D In Frail Elderly Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A9001116
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2009-01-08 (Estimated); Status verified 2009-01

CONDITIONS: Elderly, Frail
MeSH Terms: interventions — Vitamin D; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- C (Experimental)
  Interventions: Procedure: Vitamin D Placebo + Exercise
- B (Experimental)
  Interventions: Drug: Vitamin D + Sham Exercise
- A (Experimental)
  Interventions: Drug: Vitamin D + Exercise
- D (Placebo Comparator)
  Interventions: Procedure: Vitamin D Placebo + Sham Exercise

INTERVENTIONS:
Drug: Vitamin D + Sham Exercise — 1000 IU per day of Vitamin D + Sham (equivalent to placebo) Exercise
  Arms: B
Procedure: Vitamin D Placebo + Exercise — Vitamin D placebo + Exercise
  Arms: C
Procedure: Vitamin D Placebo + Sham Exercise — Vitamin D placebo + Sham (equivalent to placebo) Exercise
  Arms: D
Drug: Vitamin D + Exercise — 1000 IU per day of Vitamin D + Exercise
  Arms: A

SUMMARY:
The study will explore multiple mobility function tests as well as functional and neuropsychological tests in elderly subjects at risk for falls and disability, before and after 4-month exercise and/or Vitamin D intervention.

DETAILED DESCRIPTION:
The study was terminated on 10Jan2008. This was a strategic decision not related to safety, efficacy, or feasibility of trial.

ELIGIBILITY:
Inclusion Criteria:

* Elderly subjects with moderate frailty residing in assisted living facilities.

Exclusion Criteria:

* Presence of progressive, unstable chronic disease; hyperparathyroidism, hypercalcemia.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-10; Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Characterization of effect of 4-month exercise and/or Vitamin D intervention on mobility function and strength in frail elderly subjects. | Throughout trial

SECONDARY OUTCOMES:
Evaluation of utility and variability of mobility function tests and biomarkers, as well as explore the predictors for the exercise and/or Vitamin D intervention response in frail elderly subjects. | throughout trial

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Farmington, Connecticut
  - Pfizer Investigational Site, Hyattsville, Maryland
  - Pfizer Investigational Site, Roslindale, Massachusetts
  - Pfizer Investigational Site, New York, New York

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001116&StudyName=Randomized%20study%20of%20exercise%20and%20Vitamin%20D%20in%20Frail%20Elderly%20subjects.